CLINICAL TRIAL: NCT01710449
Title: Evaluation of Regional Ventilation in Normal Subjects and Subjects With Airway and Lung Disorders (COPD, Asthma, Emphysema, Small Airway Disease and Cystic Fibrosis) Using 19F MRI of Inert Perfluorinated Gases Mixed With Oxygen.
Brief Title: Evaluation of Regional Ventilation Using 19F MRI of Inert Perfluorinated Gases Mixed With Oxygen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hal C Charles (Other)
Responsible Party: Sponsor-Investigator, Hal C Charles, Associate Professor Department of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00015170; DIAL1001001 (Other: Duke University Medical Center)
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-11

CONDITIONS: COPD; Asthma; Cystic Fibrosis; Emphysema; Small Airways Diseases
Keywords: Lung Transplant
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Cystic Fibrosis; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal (Experimental): The subjects will receive the gas by breathing perfluorinated gas/oxygen mixture using either a disposable Mouthpiece without Bite blocks or Disposable oral-nasal (full Face) Non Invasive Ventilation with no Anti Asphyxia Vents no vent CAPA/NPPV Face mask and a standard Douglas Bag system.
  Interventions: Drug: perfluorinated gas/oxygen mixture
- Lung Disease (Experimental): The subjects will receive the gas by breathing perfluorinated gas/oxygen mixture using either a disposable Mouthpiece without Bite blocks or Disposable oral-nasal (full Face) Non Invasive Ventilation with no Anti Asphyxia Vents no vent CAPA/NPPV Face mask and a standard Douglas Bag system.
  Interventions: Drug: perfluorinated gas/oxygen mixture

INTERVENTIONS:
Drug: perfluorinated gas/oxygen mixture — Subjects are imaged with MRI one time in an proof of concept study for the use of perfluorinated gas / oxygen mixtures as an MRI contrast agent for lung function.

SUMMARY:
An open label study in 40-60 subjects with diagnosed lung airway disease and in 10-20 normal controls. Each subject will receive PFP as a contrast agent to visualize the airway and alveolar spaces in their lungs using magnetic resonance imaging of inert gas/oxygen mixtures.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the utilization of conventional 'thermally' polarized perfluorinated gas mixed with oxygen as an exogenous inert contrast agent to image the airway spaces in normal and diseased human lungs. This is an open label proof of concept study expanding on work by other groups in animals and ex-vivo human lungs and on studies in human subjects with such gases. Projection images (2-dimensional) and 3D images will be obtained using 19F MRI coupled with spirometry breathing maneuvers to correlate spirometry variables (e.g. FEV1 and FEV1/FVC) with regional distribution of the gas.

ELIGIBILITY:
Subjects with Lung and/or Airway Disease

-Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Subjects must be ≥ 18 years of age;
2. Evidence of lung disease or injury by medical history, physical exam, and/or clinical laboratories;

   1. COPD
   2. Asthma
   3. Cystic Fibrosis
   4. Emphysema/Other Small Airways Diseases
   5. Lung Transplant
3. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
4. Subjects who are willing and able to comply with scheduled visits and other trial procedures.

   * Exclusion Criteria

Subjects presenting with any of the following will not be included in the trial:

1. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
2. Unable to receive gas mixture by breathing because of contraindications;
3. Participation in a clinical trial with a study drug that may impact lung function in the past 14 days; or
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
5. Female; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Normal Subjects

-Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the trial:

1. Subjects must be ≥ 18 years of age;
2. Non-smokers;
3. No Evidence of prior lung disease or lung injury by medical history, physical exam, and/or clinical laboratories;
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the trial.
5. Subjects who are willing and able to comply with scheduled visits and other trial procedures.

   * Exclusion Criteria

Subjects presenting with any of the following will not be included in the trial:

1. Unable to undergo a 3.0-Tesla MRI exam of the lungs and chest because of contraindications (e.g. metal in the eye, claustrophobia);
2. Unable to receive gas mixture by breathing because of contraindications;
3. Participation in a clinical trial with a study drug that may impact lung function in the past 14 days; or
4. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
5. Female; women of childbearing potential must have a confirmed negative urine pregnancy test on the day of the MR scan, prior to the MRI scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
MRI image quality of Perfluorinated Gas imaging of the lung | Single exposure
  Identify Image quality characteristics related to lung function characterized by 19F MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Cecil Charles, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States